CLINICAL TRIAL: NCT01803412
Title: An Open-label Extension Study of the Long-term Safety, Tolerability and Efficacy of Drisapersen in US and Canadian Subjects With Duchenne Muscular Dystrophy.
Brief Title: A Study of the Safety, Tolerability & Efficacy of Long-term Administration of Drisapersen in US & Canadian Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMD115501
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Muscular Dystrophies
Keywords: GSK2402968; open-label extension; safety; drisapersen; Duchenne Muscular Dystrophy; tolerability; Quality of Life
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne | interventions — PRO051

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Alternate Intravenous Dosing Arm (Experimental): Subjects will receive drisapersen as a regimen of 3 mg/kg over 1 hr IV weekly throughout the duration of participation.
  Interventions: Drug: Drisapersen
- Primary continuous Dosing Arm (Experimental): Subjects will receive drisapersen 6 mg/kg as SC injection(s) once a week, continuously throughout their duration of participation.
  Interventions: Drug: Drisapersen
- Alternate Intermittent Dosing Arm (Experimental): Subjects will receive drisapersen intermittently, as a regimen of 6 mg/kg as SC injection(s) once a week for 8 weeks followed by 4 weeks of no dosing, throughout their duration of participation.
  Interventions: Drug: Drisapersen

INTERVENTIONS:
Drug: Drisapersen — Drisapersen will be supplied as 3 mL (milliliter) vials containing 1 mL sterile solution of 200 mg/mL strength. Each subject will receive drisapersen 3 mg/kg administered IV once a week, continuously throughout their duration of participation
  Other Names: BMN 051
  Arms: Alternate Intravenous Dosing Arm
Drug: Drisapersen — Drisapersen will be supplied as 3 mL (milliliter) vials containing 1 mL sterile solution of 220 mg/mL strength. Each subject will receive drisapersen 6 mg/kg administered SC once a week, either continuously or intermittently (for 8 weeks, followed by 4 weeks of no dosing) throughout their duration of participation
  Other Names: BMN 051
  Arms: Primary continuous Dosing Arm
Drug: Drisapersen — Drisapersen will be supplied as 3 mL (milliliter) vials containing 1 mL sterile solution of 220 mg/mL strength. Each subject will receive drisapersen 6 mg/kg administered SC once a week, either continuously or intermittently (for 8 weeks, followed by 4 weeks of no dosing) throughout their duration of participation
  Other Names: BMN 051
  Arms: Alternate Intermittent Dosing Arm

SUMMARY:
This is a phase III, multicenter, open-label, uncontrolled extension study in male subjects with DMD open to eligible US and Canadian subjects who previously participated in the following studies of drisapersen: DMD114876, DMD114044 and DMD114349. Subjects will receive 6mg/kg subcutaneous drisapersen on a weekly basis. For subjects who have previously experienced significant safety or tolerability issues or who experience these during the study, there is the potential of an alternate intermittent dosing arm that will be given as a regimen of 6 mg/kg weekly for 8 weeks followed by 4 weeks off treatment. For subjects who experience or have previously experienced significant safety/tolerability issues, side effects or reactions or intermittent dosing, intravenous dosing will be made available.

DETAILED DESCRIPTION:
In Part A of the study (DMD115501, original protocol), 21 subjects entered the study at 3 US sites and completed up to 14 weeks of treatment, and up to 22 weeks of follow-up. This protocol amendment, Part B of the study will include up to 13 more US and Canadian centers, and up to 51 more subjects. In total the study will enroll approximately 72 subjects. All subjects will commence Part B at screening and follow the study schedule.

The primary dosing arm is drisapersen 6 mg/kg as SC injection(s) once a week. For subjects who have previously experienced significant safety or tolerability issues or who experience these during the study, there is the potential of an alternate intermittent dosing arm that will be given as a regimen of 6 mg/kg/wk for 8 weeks followed by 4 weeks of treatment. For subjects who experience or have previously experienced significant safety/tolerability issues, intravenous dosing will be made available.

This study does not have a minimum duration of participation. Subjects will have varying times of study participation depending on when they enter from one of the eligible studies, and will be permitted to continue in this study until such a time that they withdraw based on protocol-defined criteria, or BioMarin stops the study.

ELIGIBILITY:
Inclusion Criteria:

* Participation in an eligible drisapersen study as follows:

(A) Prior DMD114876 subjects: Subjects who completed both the 24 week double-blind treatment and 24 week post-treatment phases in study DMD114876 OR Subjects who withdrew from the treatment portion of study DMD114876 due to meeting laboratory safety stopping criteria may be eligible to enrol in the extension study if: the laboratory parameters that led to stopping have resolved; the principal investigator (PI) considers the benefit of further treatment with drisapersen outweighs the risk to the individual subject; and following consultation with the Medical Monitor (B) Prior DMD114044 Subjects: US subjects who completed study DMD114044 in another country and who want to return to the US to participate in study DMD115501, upon agreement by a DMD115501 Investigator OR US citizens who participated in DMD114044 but who had to withdraw from the study due to meeting laboratory safety stopping criteria may be eligible to enrol in DMD115501 if: the laboratory parameters that led to stopping have resolved; the PI considers the benefit of further treatment with drisapersen outweighs the risk to the individual subject; and following consultation with the Medical Monitor and upon agreement by a DMD115501 investigator (C) Prior DMD114349 Subjects: US subjects who participated in and completed study DMD114044 in another country and who entered into the ongoing open-label extension study DMD114349 in a country outside the US who wish to withdraw from DMD114349 and return to the US to participate in study DMD115501, upon agreement by a DMD115501 investigator.

Canadian subjects who participated in the DMD114349 study OR Canadian subjects who withdrew from the treatment portion of the study DMD114349 due to meeting laboratory safety stopping criteria may be eligible to enroll in the extension study if the laboratory parameters that led to stopping have resolved; the PI considers the benefit of further treatment with drisapersen outweighs the risk to the individual subject; and following consultation with the Medical Monitor.

* Continued use of glucocorticoids for a minimum of 60 days prior to study entry with a reasonable expectation that the subject will remain on steroids for the duration of the study. Changes to or cessation of glucocorticoids will be at the discretion of the PI in consultation with the subject/parent and the Medical Monitor. If subject is not on steroids, involvement in the study needs to be discussed with the medical monitor.
* Willing and able to comply with all protocol requirements and procedures (with the exception of those assessments requiring a subject to be ambulant, for those subjects who have lost ambulation)
* Able to give informed assent and/or consent in writing signed by the subject and/or parent(s)/legal guardian (according to local regulations)

Exclusion Criteria:

* Subject had a serious adverse experience or who met safety stopping criteria that remains unresolved from studies DMD114876, DMD114044, or DMD114349, which in the opinion of the investigator could have been attributable to study medication, and which is ongoing. Once resolved, subject may be eligible to enrol following PI consultation with the Medical Monitor
* Use of anticoagulants, antithrombotics or antiplatelet agents, or previous treatment with investigational drugs except for drisapersen, within 28 days of the first administration of study medication
* Participation in any other investigational clinical trial within 30 days prior to the start of screening, or during this clinical study. If subject has participated in any other study within 6 months, this should be discussed with the medical monitor prior to study entry.
* History of significant medical disorder which may confound the interpretation of either efficacy or safety data (e.g. current or history of renal or liver disease/impairment, history of inflammatory illness)
* Symptomatic cardiomyopathy. If subject has a left ventricular ejection fraction <45% at Screening, the investigator should discuss inclusion of subject in the study with the medical monitor
* A platelet count under the lower limit of normal at screening. A re-test within the screening period is permissible and if within normal range the subject may enter the study.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | Up to 48 weeks
  AEs will be assessed from Pre-baseline visit until 20 weeks after the subject has either completed the study or withdrawn from treatment early. AEs are any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Systolic and diastolic blood pressure measurements to assess the safety and tolerability | Up to 48 weeks
Pulse rate and respiratory rate measurements to assess the safety and tolerability | Up to 48 weeks
Body temperature measurements to assess the safety and tolerability | Up to 48 weeks
12-Lead Electrocardiogram (ECG) measurements to assess the safety and tolerability | Up to 48 weeks
  The following parameters will be assessed: heart rate, intervals, corrected QT (QTc) interval (Bazett). In addition, an assessment of abnormal morphology will be made
Echocardiogram measurements to assess the safety and tolerability | Up to 48 weeks
  The following parameters will be assessed: Left ventricular end-diastolic/end-systolic wall thickness (septum, posterior wall), fractional shortening (SF) and ejection fraction (LVEF) will be derived from M-mode (from the parasternal long-axis or short-axis view) for quantitative measurements
Laboratory tests to assess the safety and tolerability | Up to 48 weeks
  Laboratory tests will include hematology, biochemistry and urinalysis parameters

SECONDARY OUTCOMES:
Muscle function assessment using 6-minute walking distance (6MWD) test | Up to 48 weeks
  Subjects will be asked to walk, at their own preferred speed, up and down a fixed distance until they are told to stop after 6 minutes. The subjects are warned of the time and are told that they may stop earlier if they feel unable to continue. The total distance walked within 6 minutes (or until the subject stopped in case of early termination of the test) will be recorded in meters, as well as any falls. Subjects who became non-ambulant in the prior study or who become non-ambulant during this study will not be able to perform this
North Star Ambulatory Assessment (NSAA) | Up to 48 weeks
  The NSAA is a functional scale devised from the Hammersmith Scale of Motor Ability specifically for use in ambulant children with DMD. It consists of 17 activities graded 0 (unable to perform), 1 (performs with modifications), 2 (normal movement). The scale assesses activities that are required for ambulatory activity and includes items that are rarely achieved in untreated DMD (jump, hop, raise head) as well as items that are known to progressively deteriorate over time (stand from a chair, walk)
Pulmonary function assessment | Up to 48 weeks
  Non-invasive spirometry will be conducted to determine actual and percent values for Forced Vital Capacity (FVC) and Forced Expiratory Volume (FEV1)
Time to major disease milestones | Up to 48 weeks
  Major disease milestones are defined as those events that occurred since the last time they were assessed and include the following muscular dystrophy-related milestones: Achilles tendon contracture, hamstring contracture, lumbar lordosis, limb skeletal deformity, loss of ambulation, respiratory support during the day, respiratory support during sleep, scoliosis, use of leg braces, use of orthoses, use of special shoes, using Gower's maneuver or other milestone (to be specified)
Functional Outcomes assessment | Up to 48 weeks
  One assessments will be completed to observe the changes in the ability of the subject to perform usual day-to-day activities during the study: Functional Outcomes Survey - by the family/caregivers who attends the scheduled clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: BioMarin Clinical Trials, Study Director — BioMarin Pharmaceutical
Locations (13):
- United States (10):
  - UC Davis Medical Center, Sacramento, California
  - Shriner's Hospital for Children Tampa, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Shriners Hospitals For Children, Portland, Oregon
- Canada (3):
  - Children's & Women's Health Centre of BC, Vancouver, British Columbia
  - Children's Hospital London Health Sciences Centre, London, Ontario
  - CHU Ste-Justine, Montreal, Quebec